CLINICAL TRIAL: NCT00294918
Title: Multicenter Open-label, Randomized, Dose-finding, Parallel-group, Safety and Efficacy Trial of Subcutaneous Administration of Serostim® (Mammalian Cell-derived Recombinant Human Growth Hormone, r-hGH) in the Maintenance of the Treatment Effect Obtained During the Study of Serostim® in Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS)
Brief Title: An Efficacy and Safety Trial of Serostim® in the Maintenance of the Treatment Effect Obtained During the Study of Serostim® in Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23056
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS); Human Immunodeficiency Virus Infections
Keywords: Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS); Human Immunodeficiency Virus Infections; Serostim®; recombinant human growth hormone (r-hGH)
MeSH Terms: interventions — Human Growth Hormone; Growth Hormone

ARMS (3):
- Serostim® (1 mg) (Experimental)
  Interventions: Drug: Serostim®
- Serostim® (2 mg) (Experimental)
  Interventions: Drug: Serostim®
- Serostim® (4 mg) (Experimental)
  Interventions: Drug: Serostim®

INTERVENTIONS:
Drug: Serostim® — Serostim® will be administered subcutaneously at a dose of 1 mg to subjects who had encountered toxicity during the antecedent protocol (Study 22388) whereas, other subjects will be randomized in 1:1 ratio, to receive either 2 milligram (mg) or 4 mg (on a weight adjusted basis) daily, starting from Day 1 of Week 1 up to Week 12 (Period 1). During Period 1, subjects who encounter toxicity will receive 1 mg Serostim® subcutaneously, daily for Period 2, starting from Day 1 of Week 13, whereas other subjects will be randomized in a 1:1 ratio to receive either 2 mg or 1 mg (on a weight adjusted basis) up to Week 36.
  Other Names: recombinant human growth hormone (r-hGH)

SUMMARY:
This is an open-label, multi-center, randomized, parallel-group, maintenance trial of Serostim® in subjects who have completed a prior Serostim® Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS) trial (Study 22388). The subjects, who encountered toxicity during the antecedent protocol, will be assigned to a 1 milligram (mg) dose. All other subjects will be randomized in 1:1 ratio, to receive up to 2 mg or 4 mg of Serostim®, beginning from Day 1 of Week 1. Doses will be adjusted downward in subjects weighing less than 55 kilogram (kg). Serostim® therapy will be continued at the assigned doses through Week 12 (Period 1). Subjects, who will encounter toxicity during Period 1, will be assigned to the 1 mg group for Period 2. All other subjects will be randomized in a 1:1 ratio to receive up to 2 mg or 1 mg of Serostim® on a weight adjusted basis. Period 2 therapy will begin on Day 1 of Week 13, continuing through Week 36. Study visits are required at Screening (that is, Final Visit of the antecedent trial), Day 1 of Week 1 (Baseline), and at Weeks 2, 6, 12, 14, 24, 30 and 36.

ELIGIBILITY:
Inclusion Criteria:

* Complete all treatments prescribed by the antecedent protocol (Study 22388)
* Be able and willing to comply with the protocol for the duration of the study, including concomitant therapy restrictions
* Have given written informed consent
* If female, be post-menopausal, surgically sterile, or using adequate contraception

Exclusion Criteria:

* Experienced a protocol defined toxicity or any other adverse event, which caused premature withdrawal from the antecedent study (Study 22388)
* Withdrew from the antecedent study or was discontinued prematurely for any other reason
* Based on the Final Visit evaluations from the antecedent trial, would be required to withdraw from the antecedent protocol, if (theoretically) the antecedent trial continued beyond the Final Visit
* Based on the Final Visit evaluations from the antecedent trial, would be required to temporarily stop or reduce the dose of study drug, if (theoretically) the antecedent trial continued beyond the Final Visit. This does not apply to subjects whose study drug was temporarily stopped or whose study drug dose was reduced prior to the Final Visit (Screening), provided they continued in the antecedent protocol and are stable at the time of the Final Visit (Screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2001-09; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Percent change from Week 12 in trunk fat quantified by Dual-energy X-ray absorptiometry (DXA) at Week 36 | Week 12 and Week 36

SECONDARY OUTCOMES:
Change from Week 12 in ratio of trunk fat to limb fat quantified by DXA at Week 36 | Week 12 and Week 36
Change from Week 12 in weight measured on a calibrated scale at Week 36 | Week 12 and Week 36
Change from Week 12 in total body fat quantified by DXA at Week 36 | Week 12 and Week 36
Change from Week 12 in lean body mass quantified by DXA at Week 36 | Week 12 and Week 36
Change from Week 12 in maximal chest, waist, and hip circumference at Week 36 | Week 12 and Week 36
Change from Week 12 in waist/hip ratio at Week 36 | Week 12 and Week 36
Change from Week 12 in Dorsocervical Fat Pad at Week 36 | Week 12 and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Norma Muurahainen, M.D. PhD, Study Director — EMD Serono

REFERENCES:
- [Background] Low-dose Maintenance Therapy with Recombinant Human Growth Hormone Sustains Effects of Previous r-hGH Treatment in HIV+ Patients with Excess Center Fat: Treatment Results at 60 Weeks D P Kotler, C Grunfeld, N Muurahainen, C Wanke, M Thompson, D Bock, J Gertner, and Serostim in the Treatment of Adipose Redistribution Syndrome (STARS) Trial Investigator Group. Abstract. 11th Conference on Retroviruses and Opportunistic Infections. February 8-11, 2004, Moscone West, San Francisco CA, USA.
- See also: Related Info — http://www.retroconference.org/2004/cd/Abstract/80.htm
- See also: Full FDA approved prescribing information can be found here — http://www.serostim.com